CLINICAL TRIAL: NCT00561301
Title: Biweekly Gemcitabine-Oxaliplatin and Dexamethasone for Relapsed/Refractory Malignant Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-012A
Record Dates: First submitted 2007-11-18; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention)
  Interventions: Drug: GemDOx

INTERVENTIONS:
Drug: GemDOx — gemcitabine oxliplatin

SUMMARY:
- To evaluate the feasibility of combination chemotherapies comprising of gemcitabine-dexamethasone-oxaliplatin for patients with refractory or relapsed malignant non-Hodgkin lymphoma (NHL)

DETAILED DESCRIPTION:
- The feasibility will be evaluated in terms of objective response rate, efficacy of stem cell collection, disease-free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have refractory to first-line CHOP-like regimen
* Patients who have first relapse after
* first-line CHOP-like regimen
* upfront autologous or allogeneic hematopoietic stem cell transplantation
* Age 15 years or more
* ECOG performance status ≤ 2
* Adequate bone marrow function
* Adequate kidney,liver,cardiac

Exclusion Criteria:

* Patients who have received GEM or OX

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2006-11; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 10/2009

SECONDARY OUTCOMES:
toxicities, progression-free survival, overall survival, ASCC efficacy, rate for proceeding to ASCT | 10/2009

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, professor, Principal Investigator — Ulsan Universtity Hospital, ROK
Locations (1):
- Asan Medical Center, Seoul, South Korea